CLINICAL TRIAL: NCT05895149
Title: Effects of Osteopathy in Autonomic Nervous System: a Double-blind Randomized Controlled Trial
Brief Title: Effects of Osteopathy in Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1-005
Record Dates: First submitted 2023-05-25; First posted 2023-06-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Autonomic nervous system; Heart rate variability; Osteopathy; Flying buttress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will pull from a bag within equally number of folded papers with letter 1 to 50 and it will be handled to the investigator. The even numbers correspond to the control group and the odd numbers to the experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In each participant, HRV will be measured for 2 minutes, then the flying buttress technique will be applied. After the technique, HRV will be recorded for 2 minutes, and 5 minutes later, HRV will be measured again for 2 minutes.
  Interventions: Other: Flying buttress technique
- Control group (Placebo Comparator): In each participant, HRV will be measured for 2 minutes, then the placebo technique will be applied. After the technique, HRV will be recorded for 2 minutes, and 5 minutes later, HRV will be measured again for 2 minutes.
  Interventions: Other: Placebo technique

INTERVENTIONS:
Other: Flying buttress technique — With the volunteer in a supine position, the researcher who applied the technique positioned himself standing at the head of the massage table, supporting the patient's head. He contacted the occipital region, near the occipital-mastoid suture, with the thenar and hypothenar region of his right hand. He contacted the mastoid process of the contralateral temporal bone with the thenar and hypothenar region of his left hand. The forearms were positioned in a straight line. After a slight initial compression, the researcher applied a rhythmic pumping motion with both upper limbs in a convergent direction. The pressure applied was due to the rhythmic movement of the researcher's body. The technique was performed bilaterally and each one lasted for 2 minutes
  Arms: Experimental group
Other: Placebo technique — With the volunteer in a supine position, the researcher placed the palms of their hands on the patient's shoulders. The palm of the hand rested on the acromioclavicular joint with the rest of the hand relaxed. The placebo technique was performed for 4 minutes.
  Arms: Control group

SUMMARY:
The most important regulatory system in the body is the autonomic nervous system. There are several studies that evaluate the effect of techniques applied at the base of the skull on the autonomic nervous system. The aim of this study is to evaluate the effect of the flying buttress technique on the autonomic nervous system.

DETAILED DESCRIPTION:
The most important homeostatic regulatory system in the body is the autonomic nervous system (ANS), as it coordinates functions of many organs and tissues, including the cardiac muscle.

ANS regulation in most visceral organs reflects a balance between sympathetic and parasympathetic modulation. In the neural control of the heart, there is a balance between sympathetic excitation and vagal inhibition of sinoatrial node activity, which contribute to fluctuations in heartbeat, known as heart rate variability (HRV).

HRV is considered a valuable non-invasive measurement tool for assessing ANS function, as it is relatively simple and quickly performed.

Previous studies provide evidence that osteopathic treatment is associated with changes in HRV that appear to be indicative of increased cardiac vagal modulation in various conditions.

The aim of this study is to evaluate the effect of the osteopathic technique flying buttress on the ANS through HRV.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18 and 35 years of age;
* Ability to maintain a supine position for 30 minutes;
* Healthy volunteers.

Exclusion Criteria:

* Presence of acute or chronic pain;
* Recent cranial and/or cervical injury;
* History of cranial and/or cervical surgery;
* Oncological disease;
* Brain injury;
* Cardiovascular pathology;
* Neurological pathology;
* Psychological/emotional disorder;
* Pregnancy;
* Manual therapy treatment in the last month;
* Consumption of alcohol, drugs, tobacco, chocolate, and sodas in the last 48 hours;
* Consumption of caffeine on the day of the study;
* Extreme physical exercise in the last 24 hours;
* Less than 6 hours of sleep on the night preceding the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HRV at immediately post-intervention | immediately post-intervention
  The R-R intervals will be collected using a Polar H10 chest strap (Polar Electro Oy, Kempele, Finland), and subsequently, the rMSSD and pNN50 value will be calculated using Software Kubios HRV Standard, version 3.5.0 (Biosignal Analysis and Medical Imaging Group, Department of Physics, University of Kuopio, Kuopio, Finland)
Change from baseline in HRV at 7 min post-intervention | 7 min post-intervention
  The R-R intervals will be collected using a Polar H10 chest strap (Polar Electro Oy, Kempele, Finland), and subsequently, the rMSSD and pNN50 value will be calculated using Software Kubios HRV Standard, version 3.5.0 (Biosignal Analysis and Medical Imaging Group, Department of Physics, University of Kuopio, Kuopio, Finland)

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Instituto Politécnico do Porto
Locations (1):
- Escola Superior de Saúde do Instituto Politécnico do Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arienti C, Farinola F, Ratti S, Dacco S, Fasulo L. Variations of HRV and skin conductance reveal the influence of CV4 and Rib Raising techniques on autonomic balance: A randomized controlled clinical trial. J Bodyw Mov Ther. 2020 Oct;24(4):395-401. doi: 10.1016/j.jbmt.2020.07.002. Epub 2020 Jul 31. PMID 33218540
- [Background] Cardoso-de-Mello-E-Mello-Ribeiro AP, Rodriguez-Blanco C, Riquelme-Agullo I, Heredia-Rizo AM, Ricard F, Oliva-Pascual-Vaca A. Effects of the Fourth Ventricle Compression in the Regulation of the Autonomic Nervous System: A Randomized Control Trial. Evid Based Complement Alternat Med. 2015;2015:148285. doi: 10.1155/2015/148285. Epub 2015 Jun 14. PMID 26199632
- [Background] Carnevali L, Lombardi L, Fornari M, Sgoifo A. Exploring the Effects of Osteopathic Manipulative Treatment on Autonomic Function Through the Lens of Heart Rate Variability. Front Neurosci. 2020 Oct 7;14:579365. doi: 10.3389/fnins.2020.579365. eCollection 2020. PMID 33117124
- [Background] Curi ACC, Maior Alves AS, Silva JG. Cardiac autonomic response after cranial technique of the fourth ventricle (cv4) compression in systemic hypertensive subjects. J Bodyw Mov Ther. 2018 Jul;22(3):666-672. doi: 10.1016/j.jbmt.2017.11.013. Epub 2017 Dec 9. PMID 30100295
- [Background] Gibbons CH. Basics of autonomic nervous system function. Handb Clin Neurol. 2019;160:407-418. doi: 10.1016/B978-0-444-64032-1.00027-8. PMID 31277865
- [Background] Laborde S, Mosley E, Thayer JF. Heart Rate Variability and Cardiac Vagal Tone in Psychophysiological Research - Recommendations for Experiment Planning, Data Analysis, and Data Reporting. Front Psychol. 2017 Feb 20;8:213. doi: 10.3389/fpsyg.2017.00213. eCollection 2017. PMID 28265249
- [Background] McCraty R, Shaffer F. Heart Rate Variability: New Perspectives on Physiological Mechanisms, Assessment of Self-regulatory Capacity, and Health risk. Glob Adv Health Med. 2015 Jan;4(1):46-61. doi: 10.7453/gahmj.2014.073. PMID 25694852
- [Background] Ricard, F. (2014). Tratado de Osteopatía Craneal. Articulación Temporomandibular. Análisis y tratamiento ortodóntico. (E. Medos, Ed. 3ª ed.).
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Schaffarczyk M, Rogers B, Reer R, Gronwald T. Validity of the Polar H10 Sensor for Heart Rate Variability Analysis during Resting State and Incremental Exercise in Recreational Men and Women. Sensors (Basel). 2022 Aug 30;22(17):6536. doi: 10.3390/s22176536. PMID 36081005
- [Background] Munoz ML, van Roon A, Riese H, Thio C, Oostenbroek E, Westrik I, de Geus EJ, Gansevoort R, Lefrandt J, Nolte IM, Snieder H. Validity of (Ultra-)Short Recordings for Heart Rate Variability Measurements. PLoS One. 2015 Sep 28;10(9):e0138921. doi: 10.1371/journal.pone.0138921. eCollection 2015. PMID 26414314